CLINICAL TRIAL: NCT00926796
Title: Randomized Clinical Trial Evaluating the Efficacy of Gentamicin/Azithromycin and Gemifloxacin/Azithromycin Combination Therapies as an Alternative Regimen for Uncomplicated Urogenital Gonorrhea
Brief Title: Efficacy of Combination Therapies for Gonorrhea Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-0042
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Results first posted 2014-03-20 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2013-06

CONDITIONS: Gonorrhoea
Keywords: gonorrhea, gonococcal infections, Neisseria gonorrhoeae
MeSH Terms: conditions — Gonorrhea | interventions — Azithromycin; Gentamicins; Gemifloxacin

ARMS (2):
- Regimen B: gemifloxacin plus azithromycin (Experimental): Gemifloxacin 320 mg by mouth one time plus azithromycin 2 gm by mouth one time.
  Interventions: Drug: Azithromycin; Drug: Gemifloxacin
- Regimen A: gentamicin plus azithromycin (Experimental): Gentamicin 240 mg intramuscular (IM) one time for patients greater than 45 kg or 5 mg/kg IM one time for patients less than or equal to 45 kg plus azithromycin 2 gm by mouth one time.
  Interventions: Drug: Azithromycin; Drug: Gentamicin

INTERVENTIONS:
Drug: Azithromycin — Four 500 mg tablets will be administered orally to equal a 2 gm dose.
Drug: Gentamicin — Fixed dose of 240 mg intramuscular one time for patients >45 kg and a 5 mg/kg dose for patients less than or equal to 45 kg based on their measured weight in clinic. Most patients will require 2 injections of gentamicin in separate large muscle groups.
  Arms: Regimen A: gentamicin plus azithromycin
Drug: Gemifloxacin — One 320 mg tablet administered orally.
  Arms: Regimen B: gemifloxacin plus azithromycin

SUMMARY:
The purpose of this study is to learn how to better treat gonorrhea infections. Gonorrhea is a sexually transmitted disease (STD) that is usually cured with a single antibiotic. However, some gonorrhea is not cured with a single antibiotic. The study will look at how well treating gonorrhea with 2 antibiotics works. Participants will be assigned to 1 of 2 treatment groups each receiving a combination of 2 antibiotics. Sites in the United States will recruit 500 male and female participants. Participants must be 15 to 60 years old, in good health and identified in participating sexually transmitted disease clinics as having uncomplicated cervical or urethral gonorrhea. Procedures include collection of current symptoms, medical and sexual history, sexual orientation, vital signs, height, weight, cervical/urethral cultures and clinical examinations. Volunteers will be involved for about 17 days.

DETAILED DESCRIPTION:
Infection with Neisseria (N.) gonorrhoeae carries a significant public health burden in the United States (U.S.). Gonococcal infection can result in pelvic inflammatory disease (PID), ectopic pregnancy, infertility, chronic pelvic pain, and increases the risk of transmission and acquisition of human immunodeficiency virus (HIV). With over 350,000 cases of gonorrhea reported each year, gonorrhea is the second most common notifiable condition. Furthermore, it is estimated that case reports account for only half of the incident cases of gonorrhea in the U.S. each year. Given that gonorrhea is a bacterial infection which causes symptoms in approximately 90 percent of infected men and 50 percent of infected women, the most critical aspect of reducing the public health burden of gonorrhea for affected populations is provision of effective antimicrobial therapy. In order to identify treatment options for patients with suspect or confirmed cephalosporin-resistant N. gonorrhoeae infection and patients with severe cephalosporin hypersensitivity, this study plans to determine the efficacy of each of 2 combination antimicrobial regimens for the treatment of uncomplicated gonococcal infection. This study is a multicenter clinical trial of adult males and females diagnosed with urethral or cervical gonococcal infection. Subjects will be enrolled and randomized for treatment with either Regimen A: gentamicin 240 mg intramuscular (IM) one time for patients >45 kg or 5 mg/kg IM one time for patients less than or equal to 45 kg plus azithromycin 2 gm by mouth (PO) one time, or Regimen B: gemifloxacin 320 mg PO one time plus azithromycin 2 gm PO one time. Investigators hypothesize that Regimen A will have a clinical efficacy estimate that is greater than or equal to 95 percent as well as a lower, one-sided 95 percent confidence interval (CI 95 percent) bound that is greater than or equal to 90 percent. The identical hypothesis applies for Regimen B. It should be noted that this is not a comparative trial between Regimen A and B, but rather a trial to establish efficacy data for each of these two candidate regimens. The primary objective of this study is to determine the microbiological efficacy of each of two combination antimicrobial regimens for the treatment of uncomplicated gonococcal infection (i.e., non-systemic). Secondary objectives of this study are to: assess the safety and tolerability of each candidate regimen; assess the eradication of any rectal or pharyngeal gonococcal infection by each regimen; determine the antimicrobial susceptibility profile of all gonococcal strains isolated at the time of enrollment; determine the clinical and antimicrobial susceptibility profile of all gonococcal strains isolated from patients who fail treatment; and assess the efficacy of the candidate regimens on the resolution of symptoms and signs (clinical cure). The primary efficacy analysis will be based on microbiological cure rate at end of trial based on the modified intent-to-treat (MITT) and per protocol (PP) subsets. The number, percent, and a 95 percent one-sided (lower) confidence interval of microbiological cure rate successes and failures will be computed. Additional analyses will be conducted on the following subsets: male, female, men who have sex with men (MSM) status, and subjects denying anal, oral, or vaginal intercourse during the follow-up period. Secondary endpoints will include: separate analyses of: safety and tolerability of each regimen; eradication of rectal or pharyngeal infection; antimicrobial susceptibility profile of enrollment isolates; clinical and antimicrobial susceptibility profile of treatment failures; and resolution of

ELIGIBILITY:
Inclusion Criteria:

* Male or female from 15 - 60 years old.
* Is either:

  1. Untreated male or female with urethral or cervical gonorrhea as determined by a screening laboratory test [either Nucleic Acid Amplification Test (NAAT) or culture] for Neisseria gonorrhoeae at a prior visit.
  2. Urethral or cervical gram stain demonstrating gram negative intracellular diplococci and leukocytes.
  3. Untreated male or female who is a sexual contact (anal, oral, or vaginal) of an individual with gonorrhea in the past 60 days.
* Willing to abstain from anal, oral, or vaginal sexual intercourse or use condoms until follow up is completed.
* Willing to follow up from 10 to 17 days following enrollment.
* Willing to provide written consent.
* Able to swallow pills.

Exclusion Criteria:

* Known renal insufficiency from clinical history
* Known hepatic insufficiency from clinical history
* Known QT interval prolongation from clinical history
* Known neuromuscular disorder from clinical history (i.e., myasthenia gravis or Parkinson's disease)
* Known rheumatoid arthritis or tendon disorders from clinical history
* Known kidney, heart, or lung transplants from clinical history
* Pregnant women (determined by positive urine pregnancy test)
* Breastfeeding women
* Known allergy or adverse reaction to macrolides, aminoglycosides, or quinolones
* Concomitant infection (besides chlamydia or bacterial vaginosis) which requires systemic antibiotics
* Has received systemic or intravaginal antibiotics within 30 days of study enrollment
* Currently taking corticosteroid drugs or other immunosuppressive therapy
* Currently taking cardiac antiarrhythmia drugs
* Self report of or clinical diagnosis of abdominal pain, pelvic inflammatory disease (PID), testicular pain, epididymitis, or disseminated gonococcal infection
* Self report of or clinical diagnosis of current genital ulcer (GU)
* In the judgment of the interviewer, has a medical condition or other factor that might affect their ability to follow the protocol
* Previous enrollment in this study

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 614 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Alabama Hospital - Infectious Diseases, Birmingham, Alabama
  - Los Angeles County Department of Public Health - Sexually Transmitted Disease Program, Los Angeles, California
  - San Francisco Department of Public Health - San Francisco City Clinic, San Francisco, California
  - Johns Hopkins Bayview Medical Center - Infectious Diseases, Baltimore, Maryland
  - Magee Women's Hospital of UPMC - Reproductive Infectious Disease Research, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Kirkcaldy RD, Weinstock HS, Moore PC, Philip SS, Wiesenfeld HC, Papp JR, Kerndt PR, Johnson S, Ghanem KG, Hook EW 3rd. The efficacy and safety of gentamicin plus azithromycin and gemifloxacin plus azithromycin as treatment of uncomplicated gonorrhea. Clin Infect Dis. 2014 Oct 15;59(8):1083-91. doi: 10.1093/cid/ciu521. Epub 2014 Jul 16. PMID 25031289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in outpatient STD clinics located in 5 cities across the United States.
Pre-assignment Details: Since Gonorrhea lab results were not available at randomization, participants who were found to be negative for Gonorrhea were withdrawn after randomization as they did not meet one of the eligibility criteria.
Period: Overall Study
Arm/Group | Regimen A: Gentamicin Plus Azithromycin | Regimen B: Gemifloxacin Plus Azithromycin
Started | 309 (Number randomized) | 305 (Number randomized)
Completed | 202 (Number eligible and in the full analysis set) | 199 (Number eligible and in the full analysis set)
Not Completed | 107 | 106
Not completed — Did not receive randomized treatment | 4 | 7
Not completed — Ineligible, negative for gonorrhea | 57 | 60
Not completed — Ineligible, but positive for gonorrhea | 1 | 1
Not completed — Adverse Event | 7 | 14
Not completed — Lost to Follow-up | 22 | 13
Not completed — Protocol Violation | 15 | 11
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Per protocol population. See participant flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A: Gentamicin Plus Azithromycin | Regimen B: Gemifloxacin Plus Azithromycin | Total
Number analyzed (Participants) | 202 | 199 | 401
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 3 | 9
  Between 18 and 65 years | 196 | 196 | 392
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (9.9) | 30 (9.6) | 30 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 183 | 178 | 361
Region of Enrollment [Number; unit: participants]
  United States | 202 | 199 | 401

OUTCOME MEASURES:

1. Primary Outcome: Microbiological Efficacy of Gentamicin and Azithromycin for the Treatment of Uncomplicated Gonococcal Infection
Description: Percentage of enrollees negative by culture at cervix/urethra 10-17 days after treatment, regardless of history of re-exposure, among those with positive gonococcal cultures at enrollment (microbiological cure)
Time Frame: 10-17 days after treatment.
Population: Per protocol population (all randomized participants who took study drug, positive for gonorrhea, completed follow up visit, and met additional protocol specific conditions such as key inclusion/exclusion, the 10-17 day Visit 2 window requirement, etc.)
Measure: Number; unit: percentage of participants
Arm/Group | Regimen A: Gentamicin Plus Azithromycin
Number analyzed (Participants) | 202
percentage of participants | 100
Statistical Analysis 1: Comparison: Regimen A: Gentamicin Plus Azithromycin; The null hypothesis is that the microbiological efficacy estimate (proportion of participants who are cured) is <95%; Test type: Superiority or Other; p < 0.05, Exact binomial confidence limit; If the one-sided lower 95% confidence limit is greater than 95%, the null hypothesis of the microbiological efficacy estimate is <95% is rejected; Proportion of cured participants = 100, 95% CI 1-sided [lower limit 98.53] — When the lower 95% confidence limit is >=95%, the alternative hypothesis is accepted (i.e., the microbiological cure estimate is significantly >=95%)

2. Secondary Outcome: Eradication of Rectal Infection
Description: Number of enrollees with positive rectal culture at enrollment who have negative culture 10-17 days after treatment
Time Frame: 10-17 days after treatment.
Population: Participants who were positive for rectal gonorrhea at enrollment and were in the per protocol population (all randomized participants who took study drug, positive for gonorrhea, completed follow up visit, and met additional protocol specific conditions such as key inclusion/exclusion, the 10-17 day Visit 2 window requirement, etc.)
Measure: Number; unit: participants
Arm/Group | Regimen A: Gentamicin Plus Azithromycin | Regimen B: Gemifloxacin Plus Azithromycin
Number analyzed (Participants) | 1 | 5
participants | 1 | 5

3. Secondary Outcome: Eradication of Pharyngeal Infection
Description: Number of enrollees with positive pharyngeal culture at enrollment who have negative culture 10-17 days after treatment
Time Frame: 10-17 days after treatment.
Population: Participants who were positive for pharyngeal gonorrhea at enrollment and were in the per protocol population (all randomized participants who took study drug, positive for gonorrhea, completed follow up visit, and met additional protocol specific conditions such as key inclusion/exclusion, the 10-17 day Visit 2 window requirement, etc.)
Measure: Number; unit: participants
Arm/Group | Regimen A: Gentamicin Plus Azithromycin | Regimen B: Gemifloxacin Plus Azithromycin
Number analyzed (Participants) | 10 | 15
participants | 10 | 15

4. Secondary Outcome: Antimicrobial Susceptibility Profile of Treatment Failures.
Description: For treatment failures (i.e., participants with positive culture at cervix/urethra 10-17 days after treatment), the minimum inhibitory concentrations for various antimicrobial agents (Azithromycin, Cefixime, Ceftriaxone, Ciprofloxacin, Gemifloxacin, Gentamicin, Penicillin, Tetracycline).
Time Frame: Isolates obtained at enrollment (Day 0).
Population: Participants in the per protocol population (all randomized participants who took study drug, positive for gonorrhea, completed follow up visit, and met additional protocol specific conditions such as key inclusion/exclusion, the 10-17 day Visit 2 window requirement, etc.) with treatment failure.
Measure: Median (Full Range); unit: micrograms/milliliter
Arm/Group | Regimen A: Gentamicin Plus Azithromycin | Regimen B: Gemifloxacin Plus Azithromycin
Number analyzed (Participants) | 0 | 1
micrograms/milliliter
  Azithromycin |  | 0.25 [NA to NA] — Because data was available for only 1 participant, Measure of Dispersion could not be calculated.
  Cefixime |  | 0.015 [NA to NA] — Because data was available for only 1 participant, Measure of Dispersion could not be calculated.
  Ceftriaxone |  | 0.004 [NA to NA] — Because data was available for only 1 participant, Measure of Dispersion could not be calculated.
  Ciprofloxacin |  | 0.002 [NA to NA] — Because data was available for only 1 participant, Measure of Dispersion could not be calculated.
  Gemifloxacin |  | 0.004 [NA to NA] — Because data was available for only 1 participant, Measure of Dispersion could not be calculated.
  Gentamicin |  | 4 [NA to NA] — Because data was available for only 1 participant, Measure of Dispersion could not be calculated.
  Penicillin |  | 0.5 [NA to NA] — Because data was available for only 1 participant, Measure of Dispersion could not be calculated.
  Tetracycline |  | 0.25 [NA to NA] — Because data was available for only 1 participant, Measure of Dispersion could not be calculated.

5. Secondary Outcome: Clinical Profile of Treatment Failures.
Description: For treatment failures (i.e., participants with positive culture at cervix/urethra 10-17 days after treatment), number participants with clinical symptoms (vaginal/urethral discharge, dysuria, dyspareunia) at 10-17 days.
Time Frame: 10-17 days
Population: Participants who had clinical symptoms at enrollment and were in the per protocol population (all randomized participants who took study drug, positive for gonorrhea, completed follow up visit, and met additional protocol specific conditions such as key inclusion/exclusion, the 10-17 day Visit 2 window requirement, etc.) with treatment failure.
Measure: Number; unit: participants
Arm/Group | Regimen A: Gentamicin Plus Azithromycin | Regimen B: Gemifloxacin Plus Azithromycin
Number analyzed (Participants) | 0 | 1
participants
  Vaginal/urethral discharge |  | 0
  Dysuria |  | 0
  Dyspareunia |  | 0

6. Secondary Outcome: Resolution of Symptoms and Signs (Clinical Cure)
Description: Number of participants whose gonorrhea-related symptoms (e.g. vaginal/urethral discharge, dysuria, dyspareunia) present at enrollment has resolved by visit 2.
Time Frame: 10-17 days after treatment.
Population: Participants who had clinical symptoms at enrollment and were in the per protocol population (all randomized participants who took study drug, positive for gonorrhea, completed follow up visit, and met additional protocol specific conditions such as key inclusion/exclusion, the 10-17 day Visit 2 window requirement, etc.)
Measure: Number; unit: participants
Arm/Group | Regimen A: Gentamicin Plus Azithromycin | Regimen B: Gemifloxacin Plus Azithromycin
Number analyzed (Participants) | 188 | 182
participants | 179 | 177

7. Secondary Outcome: Antimicrobial Susceptibility Profile of Enrollment Isolates.
Description: Minimum inhibitory concentration (micrograms/milliliter) of pretreatment gonorrhea isolates collected from participants
Time Frame: Isolates obtained at enrollment (Day 0).
Population: Per protocol population (all randomized participants who too study drug, positive for gonorrhea, completed follow up visit, and met additional protocol specific conditions such as key inclusion/exclusion, the 10-17 day Visit 2 window requirement, etc.).
Measure: Median (Full Range); unit: micrograms/milliliter
Groups:
- Baseline: All per protocol participants at baseline with evaluable isolates
Arm/Group | Baseline
Number analyzed (Participants) | 396
micrograms/milliliter
  Azithromycin | 0.25 [0.03 to 16]
  Cefixime | 0.015 [0.001 to 1.0]
  Ceftriaxone | 0.008 [0.001 to 0.125]
  Ciprofloxacin | 0.004 [0.002 to 32]
  Gemifloxacin | 0.004 [0.001 to 8]
  Gentamicin | 4 [0.002 to 16]
  Penicillin | 0.5 [0.004 to 64]
  Tetracycline | 0.5 [0.03 to 32]

8. Primary Outcome: Microbiological Efficacy of Gemifloxacin and Azithromycin for the Treatment of Uncomplicated Gonococcal Infection
Description: as for outcome 1
Time Frame: 10-17 days after treatment.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Regimen B: Gemifloxacin Plus Azithromycin
Number analyzed (Participants) | 199
percentage of participants | 99.50
Statistical Analysis 1: Comparison: Regimen B: Gemifloxacin Plus Azithromycin; The null hypothesis is that the microbiological efficacy estimate (proportion of participants who are cured) is <95%; Test type: Superiority or Other; p < 0.05, Exact bionomial confidence limit; [statistical method as in outcome 1, analysis 1]; Proportion of cured participants = 99.50, 95% CI 1-sided [lower limit 97.64] — When the lower 95% confidence interval is above 95%, the alternative hypothesis is accepted (i.e., the microbiological cure estimate is significantly >=95%)

9. Secondary Outcome: Number of Participants With Adverse Events for Each Regimen
Description: Number of treated participants experiencing mild, moderate, severe, or life-threatening adverse events (AEs) either temporarily associated or not associated with study product.
Time Frame: Day 0 through Day 30
Population: All participants receiving study medication comprised the safety population. Of 614 participants randomized, 603 received study medication.
Measure: Number; unit: participants
Arm/Group | Regimen A: Gentamicin Plus Azithromycin | Regimen B: Gemifloxacin Plus Azithromycin
Number analyzed (Participants) | 305 | 298
participants | 157 | 185

ADVERSE EVENTS:
Time Frame: Enrollment, at follow-up, which as targeted 10-17 days, and through 30 days.
Description: All participants who received study medication comprise the number of participants at risk.
Arm/Group | Regimen A: Gentamicin Plus Azithromycin | Regimen B: Gemifloxacin Plus Azithromycin
Serious Adverse Events (participants affected / at risk) | 0/305 | 0/298
Other Adverse Events (participants affected / at risk) | 124/305 | 164/298
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A: Gentamicin Plus Azithromycin (N=305) | Regimen B: Gemifloxacin Plus Azithromycin (N=298)
Diarrhea (Gastrointestinal disorders) | 53 (53) | 66 (67)
Nausea (Gastrointestinal disorders) | 79 (79) | 120 (121)
Vomiting (Gastrointestinal disorders) | 32 (32) | 42 (44)

LIMITATIONS AND CAVEATS:
After the SMC meeting held during August 2012, the SMC recommended halting trial enrollment because continued participant accrual to targeted enrollment of 500 infected participants would be highly unlikely to alter the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No